CLINICAL TRIAL: NCT05405556
Title: Sotagliflozin Safety and Tolerability Among Renal Transplant Recipients
Acronym: START
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martina McGrath, MD (Other)
Responsible Party: Sponsor-Investigator, Martina McGrath, MD, Associate Physician, Instructor in Medicine, Principal Investigator, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000454
Record Dates: First submitted 2022-05-20; First posted 2022-06-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Intervention Model Description: A pre-defined algorithm for suggested management of acute changes in eGFR will be provided to all treating physicians. To test the proportion of patients successfully completing the protocol according to two different eGFR reporting strategies, randomization at the patient level will occur as follows:
  1. only study-related eGFR values >25% below baseline will be reported to patients and providers
  2. all study-related eGFR values will be provided to patients and providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients and providers only aware of study eGFR values more than 25% below baseline (Experimental): Any study-related eGFR value more than 25% below the baseline measurement will be reported to the patient and treating physician.
  Interventions: Diagnostic Test: eGFR reporting
- Patients and providers aware of all study eGFR values (Other): All study-related eGFR measurements will be reported to the treating physician and patient.
  Interventions: Diagnostic Test: eGFR reporting

INTERVENTIONS:
Diagnostic Test: eGFR reporting — To test the proportion of patients successfully completing the protocol according to different eGFR reporting strategies, randomization in a 1:1 fashion at the patient level (n=50) will occur as follows:
  1. only study-related eGFR values >25% below baseline will be reported to patients and providers
  2. all study-related eGFR will be provided to patients and providers

SUMMARY:
This is an investigator-initiated, randomized controlled trial in adult KTRs (N=50) with stable allograft function to assess: 1) the reversibility of the expected acute changes in eGFR with sotagliflozin (donated by Lexicon); 2) proportion of patients completing the protocol according to different eGFR reporting strategies (using a predefined algorithm to manage the expected pharmacological effect of sotagliflozin on eGFR); 3) safety and tolerability of sotagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Recipients of kidney transplant with stable eGFR*
* eGFR-creatinine (CKD-EPI 2021) ≥25 mL/min/1.73 m2
* Informed consent

  * Stable eGFR will be ascertained by careful chart review establishing that the patient's current graft has been functioning for at least 12 months post-transplantation, patients have not been treated for acute rejection within the prior 3 months, and a creatinine-based eGFR is stable (two consecutive measurements separated by at least 28 days within 5 mL/min/1.73 m2) and ≥25 mL/min/1.73 m2.

Exclusion Criteria:

* Recurrent urinary tract infections (>2 episodes/year or antibiotic prophylaxis)
* Biopsy-proven acute rejection within 12 weeks
* Screening serum potassium >5.5 mmol/L
* Uncontrolled hypertension (systolic blood pressure >180/100 mmHg)
* New York Heart Association (NYHA) Class IV HF
* Myocardial infarction, unstable angina, revascularization procedure (e.g., stent or bypass graft surgery), or cerebrovascular accident within 12 weeks
* History of diabetic ketoacidosis
* Type 1 Diabetes Mellitus
* Hereditary glucose-galactose malabsorption or primary renal glucosuria
* Liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis); Alanine aminotransferase (ALT) levels >2.0 times the upper limit of normal (ULN) or total bilirubin >1.5 times the ULN, unless consistent with Gilbert's disease
* Malignancy within 5 years (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the cervix in situ, or a malignancy that in the opinion of the investigator is considered cured with minimal risk of recurrence)
* Human immunodeficiency virus antibody positive
* Major surgery within 12 weeks
* Atraumatic amputation within past 12 months of screening, or an active skin ulcer, osteomyelitis, gangrene, or critical ischemia of the lower extremity within 6 months of screening
* Combination use of ACEi and ARB
* Current use of an SGLT2 inhibitor (within 12 weeks prior to randomization)
* Known allergies, hypersensitivity, or intolerance to SGLT2i or its excipients
* Digoxin plasma level >1.2 ng/mL
* Clofibrate, fenofibrate, dronedarone, or ranolazine treatment that has not been at a stable dose in the 30 days prior to screening or randomization, or a dose adjustment is expected
* Received an active investigational drug (including vaccines) other than a placebo agent, or used an investigational medical device within 12 weeks before Day 1/baseline
* Pregnant or breast-feeding or planning to become pregnant or breast-feed during the study
* Women of childbearing potential not willing to use a highly-effective method(s) of birth control, or who are unwilling or unable to be tested for pregnancy
* Any condition that in the opinion of the investigator would make participation not in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Reversibility of eGFR changes | 16 weeks total
  Following 12 weeks of open-label drug treatment, participants will stop drug and be followed for a further four weeks (16 weeks total). Reversibility will be assessed as the proportion of patients who return to baseline eGFR (+/- 10%) by the end of the 4-week off-treatment period.

SECONDARY OUTCOMES:
Proportion of patients successfully completing the full treatment protocol, according to randomized groups | 16 weeks total
  Following 12 weeks of open-label drug treatment, participants will stop drug and be followed for a further four weeks. The proportion of patients completing the full 16 weeks will be compared according to randomized groups.

OTHER OUTCOMES:
Safety Assessments | 4 weeks
  - Acute changes in eGFR (baseline to 4 weeks)
Safety Assessments | 12 weeks
  - Longer-term changes in eGFR (baseline to 12 weeks and 4 weeks to 12 weeks)
Safety Assessments | Weeks 12-16 (off-drug)
  - Reversibility of changes in eGFR (12 to 16 weeks - after drug discontinuation)
Safety Assessments | 12 weeks
  - Acute Kidney Injury (>50% increase in serum creatinine/40% decline in eGFR within one week), which will be assessed throughout the on-drug period of 12 weeks
Safety Assessments | 12 weeks
  - All adverse events (AEs)
Safety Assessments | 12 weeks
  - All serious adverse events (SAEs)
Safety Assessments | 12 weeks
  - Diarrhea
Safety Assessments | 12 weeks
  - Infection requiring treatment with anti-microbials (including urogenital infection and urinary tract infections)
Safety Assessments | 12 weeks
  - Severe hypoglycemia (event that requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions)
Safety Assessments | 12 weeks
  - Diabetic ketoacidosis
Safety Assessments | 12 weeks
  - Hyperkalemia (>5.5 mmol/L)
Safety Assessments | 12 weeks
  - Hypotension (symptomatic SBP <90 mmHg or hypotension requiring adjustment in blood pressure medications or treatment in an emergency or hospitalized setting)
Tolerability Assessments | 12 weeks
  - Proportion of participants able to complete the full 12 weeks of treatment, according to randomized arm
Tolerability Assessments | 12 weeks
  - Study medication discontinuation rates
Tolerability Assessments | 12 weeks
  - KDQOL-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martina M McGrath, MBBCh, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only sharing of anonymized data will be considered as per approved protocol. Written requests for data sharing will be considered on a case-by-case basis from qualified external researchers, based on scientific merit.

REFERENCES:
- [Background] Bhatt DL, Szarek M, Pitt B, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Inzucchi SE, Kosiborod MN, Cherney DZI, Dwyer JP, Scirica BM, Bailey CJ, Diaz R, Ray KK, Udell JA, Lopes RD, Lapuerta P, Steg PG; SCORED Investigators. Sotagliflozin in Patients with Diabetes and Chronic Kidney Disease. N Engl J Med. 2021 Jan 14;384(2):129-139. doi: 10.1056/NEJMoa2030186. Epub 2020 Nov 16. PMID 33200891